CLINICAL TRIAL: NCT07305948
Title: Prospective Evaluation of a Free Induction Decay (FID) Navigator-Based Off-Resonance Correction Method (DORK) for Improving High-Resolution 3D Echo Planar (EPI) Susceptibility-Weighted (SWI) Brain MRI
Brief Title: Evaluation of a New MRI Technique to Reduce Breathing-Related Artifacts in Brain Imaging
Acronym: DORK
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Other Study IDs: K2025-9116
Record Dates: First submitted 2025-11-27; First posted 2025-12-26 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-11

CONDITIONS: Brain Diseases
MeSH Terms: conditions — Brain Diseases | interventions — Echo-Planar Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Undergoing Routine Clinical Brain MRI
  Interventions: Diagnostic Test: Dual Free Induction Decay (FID) Navigator Off-Resonance Corrected (DORK) 3D Susceptibility Weighted (SWI) Echo Planar Imaging (EPI)

INTERVENTIONS:
Diagnostic Test: Dual Free Induction Decay (FID) Navigator Off-Resonance Corrected (DORK) 3D Susceptibility Weighted (SWI) Echo Planar Imaging (EPI) — This intervention consists of a modified magnetic resonance imaging (MRI) acquisition and reconstruction method used during routine clinical brain imaging. The method adds two very short free-induction-decay (FID) navigator signals to each repetition of a high-resolution 3D echo planar imaging (EPI) susceptibility-weighted imaging (SWI) sequence. These navigator signals measure breathing-related magnetic field changes, which are then used to perform dynamic off-resonance correction (DORK) during image reconstruction. The modified sequence does not change the clinical scan time or affect patient care. For each participant, both uncorrected and corrected SWI images are generated from the same raw data.

SUMMARY:
This study aims to improve the quality of brain magnetic resonance imaging (MRI) scans by testing a new imaging method that reduces distortions caused by breathing. During respiration, small movements of the chest and diaphragm can lead to subtle changes in the magnetic field within the head. These changes can introduce artifacts in certain MRI techniques, particularly susceptibility-weighted imaging (SWI), which is used to visualize veins, small hemorrhages, and iron deposits.

The investigated method measures breathing-related magnetic field variations during MRI acquisition using two very short navigator signals, referred to as free induction decay (FID) navigators. These signals are used to perform dynamic off-resonance correction during image reconstruction, reducing image blurring and distortion. The method does not increase scan time and does not affect standard clinical imaging.

In this study, patients scheduled for routine clinical brain MRI are asked to provide informed consent for use of their raw MRI data for research purposes. For each participant, two sets of SWI images are generated from the same acquisition: one using standard reconstruction and one using the free induction decay navigator-based dynamic off-resonance correction method (FID-DORK). The objective is to assess whether the corrected images provide improved image quality and diagnostic reliability.

The study includes adult patients undergoing routine clinical MRI at Karolinska University Hospital. Image quality is evaluated using both visual assessment by neuroradiologists and quantitative measures of image variation. No additional imaging procedures, contrast agents, or scan time are required. All research data are pseudonymized prior to analysis.

The hypothesis is that the dual free induction decay navigator-based correction method (FID-DORK) improves the diagnostic quality of high-resolution three-dimensional echo-planar imaging susceptibility-weighted imaging brain MRI by reducing breathing-related artifacts.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older)
* Undergoing a routine clinical brain MRI at Karolinska University Hospital
* Able to understand the study information and provide written informed consent
* Sequence parameters and scan protocol compatible with the research acquisition (3D-EPI SWI)

Exclusion Criteria:

* Patients unable to give informed consent
* Standard contraindications to MRI (e.g., non-MRI safe implants, severe claustrophobia)
* Clinical conditions requiring urgent imaging where research consent is not feasible
* Significant motion or incomplete scans preventing creation of research images (rare)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from adult patients referred for routine clinical brain MRI examinations at Karolinska University Hospital in Stockholm, Sweden. These individuals represent a typical clinical population undergoing MRI for a wide range of neurological indications, including tumors, vascular disorders, inflammatory conditions, and other brain diseases. Only patients scheduled for standard-of-care brain MRI that includes a susceptibility-weighted sequence (SWI) will be approached for participation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Susceptibility-Weighted Imaging Image Quality With and Without Free Induction Decay Navigator-Based Dynamic Off-Resonance Correction (FID-DORK) | Periprocedural (during the clinical brain MRI examination)
  Image quality of susceptibility-weighted imaging scans reconstructed with and without free induction decay navigator-based dynamic off-resonance correction is compared. Image quality is assessed using visual ratings by neuroradiologists and quantitative measures of image variation. Differences in image quality between corrected and uncorrected reconstructions are evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No